CLINICAL TRIAL: NCT06457178
Title: Investigation of the Effect of Acceptance and Commitment Therapy-Based Intervention on Psychological Distress and Reintegration Into Normal Life in Oncology Patients
Brief Title: Investigation of the Effect of Acceptance and Commitment Therapy-Based Intervention in Oncology Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Dilara Sert Kasım, Doctorate Student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IstanbulUC-DSKasım-001
Record Dates: First submitted 2024-05-17; First posted 2024-06-13 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acceptance and Commitment Therapy Based Intervention for Oncology Patients (Experimental): Group 1 will participate in a 5-session Acceptance and Commitment Therapy-Based Intervention for Oncology Patients intervention program.
  Interventions: Behavioral: Acceptance and Commitment Therapy-Based Intervention for Oncology Patients
- Psychoeducation for Oncology Patients (Active Comparator): Group 2 will participate in a 5-session Psychoeducation for Oncology Patients program.
  Interventions: Behavioral: Psychoeducation for Oncology Patients
- Routine Care (No Intervention): During this period, participants in group 3 will continue their routine treatment.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy-Based Intervention for Oncology Patients — An intervention program was prepared for oncology patients aiming to reduce psychological distress and increase participation in normal life.
  Arms: Acceptance and Commitment Therapy Based Intervention for Oncology Patients
Behavioral: Psychoeducation for Oncology Patients — A program was prepared to support oncology patients in physical and psychological symptom management.
  Arms: Psychoeducation for Oncology Patients

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness of Acceptance and Commitment Therapy Based Intervention for Oncology Patients. The main questions it aims to answer are:

* Does the Acceptance and Commitment to Therapy-Based Intervention for Oncology Patients affect the level of psychological distress?
* Does the Acceptance and Commitment to Therapy-Based Intervention for Oncology Patients affect the level of reintegration into normal life?

Researchers will compare Acceptance and Commitment Therapy-Based Intervention for Oncology Patients (ACT) to Psychoeducation for Oncology Patients and routine care (with no specific intervention) to see if Acceptance and Commitment Therapy-Based Intervention for Oncology Patients is effective in psychological distress and reintegration into normal living.

DETAILED DESCRIPTION:
Participants:

* They will be randomly divided into three groups (Group 1: ACT, Group 2: Psychoeducation, Group 3: Routine care).
* All participants will be asked to complete data collection forms.
* Group 1 will participate in a 5-session Acceptance and Commitment Therapy-Based Intervention for Oncology Patients intervention program.
* Group 2 will participate in a 5-session Psychoeducation for Oncology Patients program.
* During this period, participants in group 3 will continue their routine treatment.
* After completion of the interventions, participants will be asked to complete the data collection forms again.
* The researchers will then analyze the results and write the report.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Being able to read and write,
* Receiving oncologic treatment,
* Being diagnosed with breast cancer,
* To know about Medical Diagnosis,
* Being in stage 1, 2 or 3 of the disease,
* Receiving outpatient chemotherapy treatment only,
* Internet access and computer skills to participate in online group interviews,
* Low to moderate scores on the brief psychological resilience scale,

Exclusion Criteria:

* Having serious psychiatric or cognitive impairments that limit adherence to group sessions,
* Having a physical disability that may make it difficult to participate in group sessions,
* Failure to attend sessions regularly and absenteeism,
* Currently being in a psychoeducation/psychotherapy group

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
The Distress Thermometer (DT) | 1 day before intervention start
  The scale was developed to measure psychological distress in cancer patients. The problems in the list are grouped into five areas. These are daily life problems, family problems, emotional problems, faith-related problems, and physical problems. The patient marks which one or which areas of the list he/she has experienced problems in the last week. The cut-off point of the scale in our country was found to be 4. The National Comprehensive Cancer Network (NCCN) argues that patients who score 5 or above on the distress thermometer are in significant distress and should be supported by professionals.
The Distress Thermometer (DT) | through study completion, an average of 1 year
  The scale was developed to measure psychological distress in cancer patients. The problems in the list are grouped into five areas. These are daily life problems, family problems, emotional problems, faith-related problems, and physical problems. The patient marks which one or which areas of the list he/she has experienced problems in the last week. The cut-off point of the scale in our country was found to be 4. The National Comprehensive Cancer Network (NCCN) argues that patients who score 5 or above on the distress thermometer are in significant distress and should be supported by professionals.
The Distress Thermometer (DT) | one month after the end of the interventions
  The scale was developed to measure psychological distress in cancer patients. The problems in the list are grouped into five areas. These are daily life problems, family problems, emotional problems, faith-related problems, and physical problems. The patient marks which one or which areas of the list he/she has experienced problems in the last week. The cut-off point of the scale in our country was found to be 4. The National Comprehensive Cancer Network (NCCN) argues that patients who score 5 or above on the distress thermometer are in significant distress and should be supported by professionals.

SECONDARY OUTCOMES:
Reintegration to Normal Living Index (RNLI) | 1 day before intervention start
  The Reintegration to Normal Living Index (RNLI) has two sub-dimensions. These are: daily functions and self-perceptions. The scale is scored on a five-point Likert scale: Strongly Disagree (1 point), Disagree (2 points), Undecided (3 points), Agree (4 points) and Strongly Agree (5 points). Scores that can be obtained from the scale vary between 11 and 55. A high score on the scale indicates a better level of participation in normal life.
Reintegration to Normal Living Index (RNLI) | through study completion, an average of 1 year
  The Reintegration to Normal Living Index (RNLI) has two sub-dimensions. These are: daily functions and self-perceptions. The scale is scored on a five-point Likert scale: Strongly Disagree (1 point), Disagree (2 points), Undecided (3 points), Agree (4 points) and Strongly Agree (5 points). Scores that can be obtained from the scale vary between 11 and 55. A high score on the scale indicates a better level of participation in normal life.
Reintegration to Normal Living Index (RNLI) | one month after the end of the interventions
  The Reintegration to Normal Living Index (RNLI) has two sub-dimensions. These are: daily functions and self-perceptions. The scale is scored on a five-point Likert scale: Strongly Disagree (1 point), Disagree (2 points), Undecided (3 points), Agree (4 points) and Strongly Agree (5 points). Scores that can be obtained from the scale vary between 11 and 55. A high score on the scale indicates a better level of participation in normal life.

CONTACTS AND LOCATIONS:
Overall Officials: Dilara Sert Kasım, M.Sc., Principal Investigator — Istanbul University - Cerrahpasa; Hülya Bilgin, Ph.D., Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Acibadem Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No